CLINICAL TRIAL: NCT01098968
Title: Effects of a Physical Education Program Focused on Improving Physical Fitness in Adolescents Aged 12-14 Years
Brief Title: Education and Fitness: EDUFIT Study
Acronym: EDUFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Francisco B. Ortega, Post Doct Fellow, University of Granada, Department of Physiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EDUFIT
Record Dates: First submitted 2010-04-02; First posted 2010-04-05 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Physical Fitness; Body Composition; Lipid Metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal PE (No Intervention): 2 Physical Education sessions / week
- PE Volume (Experimental): 4 Physical Education sessions/week (increased volume)
  Interventions: Behavioral: Physical activity program
- PE Volume + Intensity (Experimental): 4 Physical Education sessions/week of high intensity (increased volume and intensity)
  Interventions: Behavioral: Physical activity program

INTERVENTIONS:
Behavioral: Physical activity program — School intervention program specifically designed to increase health-related physical fitness
  Arms: PE Volume; PE Volume + Intensity

SUMMARY:
EDUFIT is a group-Randomized Controlled Trial specifically designed to enhance physical fitness and other health-related factors in a school setting in adolescents.

DETAILED DESCRIPTION:
Physical fitness is a powerful marker of cardiovascular health already at early stages in life. To promote physical fitness enhancement from the school is therefore needed and this is the main aim of the EDUFIT study (EDUcation for FITness).

The participants were randomly allocated to control group (CG), experimental group 1 (EG1) and experimental group 2 (EG2). The CG received 2 physical education sessions/week, the EG1 received 4 physical education sessions/week (volume increased) and the EG2 received 4 physical education sessions/week of high intensity (volume+intensity increased). Several health-related parameters were assessed before and after a 16-weeks intervention: physical fitness (primary outcome), body composition (secondary), and lipid-metabolic profile, ventilatory parameters, blood pressure, and cognitive and academic performance (tertiary outcomes).

The hypothesis of the EDUFIT project was that to double the number of physical education classes will improve physical fitness in adolescents. The confirmation of the hypothesis could have important public health implications.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents enrolled in the Spanish Educational System, free of any muscle-skeletal problem not allowing take part in Physical Education lessons or fitness testing.

Exclusion Criteria:

* Clinical diagnosis of diabetes
* Pregnancy
* Drugs/alcohol abuse
* In general, any chronic disease that does not permit the person to perform exercise and physical education lessons.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2007-01; Primary Completion 2007-06 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Health-related physical fitness | 4 months
  Cardiorespiratory fitness; musculoskeletal fitness; motor fitness.

SECONDARY OUTCOMES:
Cardiovascular disease risk factors | 4 months
  Body composition; lipid-metabolic profile; blood pressure; ventilatory parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco B Ortega Porcel, PhD, Principal Investigator — University of Granada (Spain)
Locations (2):
- Spain (2):
  - University of Granada, Granada, Granada
  - IES Alcántara (Consejería de Educación, Formación y Empleo de la Región de Murcia), Alcantarilla, Murcia

REFERENCES:
- [Background] Ortega FB, Ruiz JR, Castillo MJ, Moreno LA, Gonzalez-Gross M, Warnberg J, Gutierrez A; Grupo AVENA. [Low level of physical fitness in Spanish adolescents. Relevance for future cardiovascular health (AVENA study)]. Rev Esp Cardiol. 2005 Aug;58(8):898-909. Spanish. PMID 16053823
- [Background] Ortega FB, Ruiz JR, Hurtig-Wennlof A, Sjostrom M. [Physically active adolescents are more likely to have a healthier cardiovascular fitness level independently of their adiposity status. The European youth heart study]. Rev Esp Cardiol. 2008 Feb;61(2):123-9. Spanish. PMID 18364180
- [Background] Ortega FB, Ruiz JR, Castillo MJ, Sjostrom M. Physical fitness in childhood and adolescence: a powerful marker of health. Int J Obes (Lond). 2008 Jan;32(1):1-11. doi: 10.1038/sj.ijo.0803774. Epub 2007 Dec 4. PMID 18043605
- [Background] Ruiz JR, Castro-Pinero J, Artero EG, Ortega FB, Sjostrom M, Suni J, Castillo MJ. Predictive validity of health-related fitness in youth: a systematic review. Br J Sports Med. 2009 Dec;43(12):909-23. doi: 10.1136/bjsm.2008.056499. Epub 2009 Jan 21. PMID 19158130
- [Background] Ortega FB, Artero EG, Ruiz JR, Vicente-Rodriguez G, Bergman P, Hagstromer M, Ottevaere C, Nagy E, Konsta O, Rey-Lopez JP, Polito A, Dietrich S, Plada M, Beghin L, Manios Y, Sjostrom M, Castillo MJ; HELENA Study Group. Reliability of health-related physical fitness tests in European adolescents. The HELENA Study. Int J Obes (Lond). 2008 Nov;32 Suppl 5:S49-57. doi: 10.1038/ijo.2008.183. PMID 19011654
- [Background] Ortega FB, Artero EG, Ruiz JR, Espana-Romero V, Jimenez-Pavon D, Vicente-Rodriguez G, Moreno LA, Manios Y, Beghin L, Ottevaere C, Ciarapica D, Sarri K, Dietrich S, Blair SN, Kersting M, Molnar D, Gonzalez-Gross M, Gutierrez A, Sjostrom M, Castillo MJ; HELENA study. Physical fitness levels among European adolescents: the HELENA study. Br J Sports Med. 2011 Jan;45(1):20-9. doi: 10.1136/bjsm.2009.062679. Epub 2009 Aug 20. PMID 19700434
- [Result] Ardoy DN, Fernandez-Rodriguez JM, Chillon P, Artero EG, Espana-Romero V, Jimenez-Pavon D, Ruiz JR, Guirado-Escamez C, Castillo MJ, Ortega FB. [Physical fitness enhancement through education, EDUFIT study: background, design, methodology and dropout analysis]. Rev Esp Salud Publica. 2010 Mar-Apr;84(2):151-68. doi: 10.1590/s1135-57272010000200004. Spanish. PMID 20571717
- See also: Official website of the HELENA Study, an European-funded project in which this research group is actively involved — http://www.helenastudy.com/
- See also: Official website of the EFFECTS-262 Research Group (University of Granada, Spain) — http://www.ugr.es/~cts262/index.html